CLINICAL TRIAL: NCT04782908
Title: Hemodynamic Characterisation of Patients Undergoing Transcatheter Tricuspid Valve Edge-to-edge Repair in Patients With Severe Tricuspid Regurgitation and Heart Failure With Preserved Ejection Fraction
Brief Title: Hemodynamic Implications of Transcatheter Tricuspid Valve Repair in HFpEF Patients
Acronym: HERACLES-HFpEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Philipp Lurz, Professor, Managing Senior Physician, Heart Center Leipzig - University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HERACLES-HFpEF
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Congestive Heart Failure; Tricuspid Regurgitation
Keywords: Heart failure with preserved ejection fraction; tricuspid regurgitation; transcatheter tricuspid valve edge-to-edge repair
MeSH Terms: conditions — Heart Failure; Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients undergoing transcatheter tricuspid valve edge-to-edge repair will undergo multimodal cardiovascular diagnostics before and after tricuspid valve repair including pressure volume loop analysis and cardiac magnetic resonance imaging
Masking Description: Outcome assessors will be blinded whether they are analysing pre or post transcatheter tricuspid valve edge-to-edge repair data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcatheter tricuspid valve edge-to-edge repair (Experimental): Patients will undergo transcatheter tricuspid valve edge-to-edge repair (TTVR) and hemodynamic characteristics will be analysed on a multimodal approach using cardiac magnetic resonance imaging and pressure volume loop analysis before and after TTVR.
  Interventions: Device: Transcatheter tricuspid valve edge-to-edge repair

INTERVENTIONS:
Device: Transcatheter tricuspid valve edge-to-edge repair — Transcatheter tricuspid valve edge-to-edge repair is an interventional approach to treat severe tricuspid regurgitation. Under general anesthesia a clip delivery system is forwarded through the vena femoralis and right atrium in the right ventricle. A clip is deployed to clamp the tricuspid valve and reduce tricuspid valve regurgitation.

SUMMARY:
The aim of the study is to investigate the pathophysiological implications of transcatheter tricuspid valve edge-to-edge repair in patient with heart failure and preserved ejection fraction and severe tricuspid regurgitation. Changes in right- and left-ventricular function as well as the interventricular dependence will be analysed on a multimodal basis including pressure-volume loop analysis and cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Severe tricuspid regurgitation with need for interventional treatment approach as decided by an interdisciplinary heart team.
* Signs and symptoms of left-sided heart failure.
* Left-ventricular ejection fraction ≥50%
* Invasive evidence of elevated left-ventricular fillings pressures (pulmonary capillary wedge pressure [PCWP] or left-ventricular end-diastolic pressure ≥15 mmHg)

Exclusion Criteria:

* Concomitant relevant mitral valve regurgitation with need for concomitant interventional treatment
* Moderate aortic stenosis.
* Pregnancy
* Contraindication to perform cardiac magnetic resonance imaging.
* Conditions rendering patient unable to give informed consent to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Periprocedural change in enddiastolic pressure volume relationship of the left ventricle | Periprocedural.
  Change in the ratio of pressure to volume of the left ventricle before and after TTVR. Measurement will take place during TTVR with patient in general anesthesia. Measures will be made using a commercially available conductance catheter. Data analysis will be performed offline using a dedicated software.

SECONDARY OUTCOMES:
Change in the estimated left ventricular end diastolic volume at 10 mmHg as estimated by the left ventricular pressure volume relationship (LVEDPVR) | Periprocedural.
  Measurement will take place during TTVR with patient in general anesthesia. Measures will be made using a commercially available conductance catheter. Data analysis will be performed offline using a dedicated software.
Change in the ratio of isovolumetric relaxation constant "Tau" and duration of diastole of the left ventricle. | Periprocedural.
  Measurement will take place during TTVR with patient in general anesthesia. Measures will be made using a commercially available conductance catheter. Data analysis will be performed offline using a dedicated software.
Change in dPdtmin | Periprocedural.
  Measurement will take place during TTVR with patient in general anesthesia. Measures will be made using a commercially available conductance catheter. Data analysis will be performed offline using a dedicated software.
Change in the early diastolic filling pattern as assessed by MRI. | Baseline and 1-month follow-up following TTVR.
  All patients will receive MRI before and 1-month after TTVR on a 1.5 tesla scanner.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Centre at University Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be made available on reasonable cooperation request.